CLINICAL TRIAL: NCT05646654
Title: Interscalene Block Versus Erector Spinae Plane Block for Shoulder Arthroscopy Anesthesia: A Randomized Controlled Trial
Brief Title: Interscalene Block Versus Erector Spinae Plane Block for Shoulder Arthroscopy Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Islam Morsy, Lecturer of Anesthesia, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35914/10/22
Record Dates: First submitted 2022-12-04; First posted 2022-12-12 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Interscalene Block; Erector Spinae Plane Block; Arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Active Comparator): 3ml lidocaine 2% will be used to anesthetize the skin. Using a 20-gauge block needle put in-plane in a cephalad-to-caudad orientation to position the tip into the fascial plane on the deep (anterior) side of the erector spinae muscle, 20 ml bupivacaine 0.5% will be injected.
  Interventions: Procedure: Erector spinae plane block
- Interscalene group (Active Comparator): Using a lateral-to-medial approach, the 25-gauge needle will be inserted into the middle scalene muscle, advanced, and placed immediately lateral to the nerve roots. the needle will be visualize using an ultrasound beam to avoid intraneural and intravascular injections. After confirming negative blood aspiration, we will inject 15 mL of 0.5% bupivacaine around the nerve roots
  Interventions: Procedure: Interscalene brachial plexus block

INTERVENTIONS:
Procedure: Erector spinae plane block — Using a 20-gauge block needle put in-plane in a cephalad-to-caudad orientation to position the tip into the fascial plane on the deep (anterior) side of the erector spinae muscle, 20 ml bupivacaine 0.5% will be injected
  Arms: Erector spinae plane block group
Procedure: Interscalene brachial plexus block — Using a lateral-to-medial approach, the 25-gauge needle will be inserted into the middle scalene muscle, advanced, and placed immediately lateral to the nerve roots. the needle will be visualize using an ultrasound beam to avoid intraneural and intravascular injections. After confirming negative blood aspiration, we will inject 15 mL of 0.5% bupivacaine around the nerve roots
  Arms: Interscalene group

SUMMARY:
The aim of this study is to compare the effectiveness of ESPB versus ISB in anesthesia for shoulder arthroscopy

DETAILED DESCRIPTION:
Regional anesthetic techniques can control pain effectively, both at rest and on movement, allowing earlier mobilization without the adverse effects of opioids. Among the various types of regional anesthetic techniques, the interscalene brachial plexus block (ISB) is a gold standard used nerve block technique for postoperative analgesia in patients undergoing shoulder surgery, as it has consistently been shown to significantly control.

the interscalene brachial plexus block (ISB) regional anesthesia offers many advantages over general anesthesia for both arthroscopic and open surgeries of the shoulder it provides excellent intraoperative anesthesia and muscle relaxation' as well as analgesia that continues into the postoperative period

ELIGIBILITY:
Inclusion Criteria:

* Patients with Body Mass Index < 40 kg/m2
* American Society of Anesthesiologists (ASA) physical status I-II
* scheduled for elective shoulder arthroscopy

Exclusion Criteria:

* Known allergy to local anesthetics
* Allergy to all opioid medications
* Diagnostic shoulder arthroscopic procedures
* Patients with chronic opioids
* Patients who converted to general anesthesia use and coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative fentanyl consumption | 30 minutes
  Fntanyl will be administered 1 µg/kg IV increments.

SECONDARY OUTCOMES:
Postoperative pain | 24 hours postoperative
  numeric rating scale (NRS) (0 represents "no pain" while 10 represents "the worst pain imaginable").
Rescue analgesia in the form of IV meperidine (0.5 mg/kg) boluses if NRS >3. Time to the 1st rescue analgesic request will be recorded | 24 hours postoperative
Total amount of rescue analgesic | 24 hours postoperative
  Rescue analgesia in the form of IV meperidine (0.5 mg/kg) boluses if NRS >3.

CONTACTS AND LOCATIONS:
Locations (1):
- Islam Morsy, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For one year after completion of the study